CLINICAL TRIAL: NCT04681417
Title: Ocular Conservative Treatment for Retinoblastoma: Efficacy of the New Management Strategies and Visual Outcome - RETINO 2018
Brief Title: Ocular Conservative Treatment for Retinoblastoma : Efficacy of the New Management Strategies and Visual Outcome
Acronym: RETINO 2018
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Fondation Rothschild Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC 2019-05
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Retinoblastoma
Keywords: Pediatric; Ocular conservative treatment in retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Melphalan; Topotecan; Etoposide; Carboplatin; Vincristine; Drug Therapy; Platinum Compounds; Hyperthermia, Induced; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study 1: Melphalan or Melphalan + Topotecan (Experimental): Randomized phase-II study evaluating the efficacy of Intra-Arterial Chemotherapy (IAC) with melphalan and topotecan versus melphalan alone, both in association with ophthalmologic treatments.
  Interventions: Drug: Melphalan or Melphalan + Topotecan; Device: Thermotherapy (local treatment); Device: Cryotherapy (local treatment); Device: Iodine-125 plaques (local treatment); Drug: Intravitreal Melphalan chemotherapy injections (local treatment)
- Study 2: Etoposide, carboplatin and vincristine (Other): Neoadjuvant chemotherapy involves 2 to 6 cycles of combined etoposide, carboplatin and vincristine in association with ophthalmologic treatments.
  Interventions: Drug: etoposide, carboplatin and vincristine or local ophthalmological treatment without IV chemotherapy; Drug: Carboplatin administered on Day 1; Device: Thermotherapy (local treatment); Device: Cryotherapy (local treatment); Device: Iodine-125 plaques (local treatment); Drug: Intravitreal Melphalan chemotherapy injections (local treatment)

INTERVENTIONS:
Drug: Melphalan or Melphalan + Topotecan — IAC: 2-6 cycles every 1 month (number based on the local tumor evolution), performed using radio-guided catheterization and delivery at the ostium of the ophthalmic artery, in neuroradiology operating room, and under General Anesthesia (GA). IAC will be administered at the Fondation Rothschild Hospital in collaboration with the Interventional Neuroradiology team.
  Other Names: Alkeran, Topotecan Accord; Topotecan Hospira chemotherapy
  Arms: Study 1: Melphalan or Melphalan + Topotecan
Drug: etoposide, carboplatin and vincristine or local ophthalmological treatment without IV chemotherapy — 2 to 6 cycles of combined etoposide, carboplatin and vincristine or local ophthalmological treatment without IV chemotherapy : thermotherapy and/or cryotherapy and/or iodine-125 plaques and/or intravitreal chemotherapy injections
  Other Names: etoposide, carboplatin and vincristine chemotherapy
  Arms: Study 2: Etoposide, carboplatin and vincristine
Drug: Carboplatin administered on Day 1 — Chemothermotherapy : Intravenous injection by carboplatin
  Other Names: platinum-based chemotherapy
  Arms: Study 2: Etoposide, carboplatin and vincristine
Device: Thermotherapy (local treatment) — Thermotherapy after carboplatin administered on Day 1
  Other Names: Thermotherapy after carboplatin administered on Day 1
Device: Cryotherapy (local treatment) — Cryotherapy (local treatment)
Device: Iodine-125 plaques (local treatment) — Iodine-125 plaques (local treatment)
Drug: Intravitreal Melphalan chemotherapy injections (local treatment) — Intravitreal Melphalan chemotherapy injections (local treatment)

SUMMARY:
This protocol includes 2 independent studies. Both studies are multicenter studies, evaluating different therapeutic approaches in two different populations of patients:

* Study 1, a randomized phase-II study evaluating the efficacy of Intra-Arterial Chemotherapy (IAC) with melphalan and topotecan versus melphalan alone, both in association with ophthalmologic treatments.
* Study 2, a minimally invasive interventional study evaluating the results on visual function following reference treatment with intravenous (IV) chemotherapy in association with ophthalmologic or local ophthalmological treatment without IV chemotherapy.

DETAILED DESCRIPTION:
Primary objective of the studies:

* Study 1: To evaluate the efficacy of IAC in term of local control of the disease in patients eligible for IAC (randomized phase II study);
* Study 2: To assess the visual function, based on World Health Organization (WHO) criteria, in patients eligible for other conservative treatments (IV chemotherapy in association with local ophthalmologic trématent or local ophthalmological treatment without IV chemotherapy; this is a minimally invasive interventional study).

ELIGIBILITY:
Inclusion Criteria:

Overall study inclusion criteria:

1. Newly diagnosed retinoblastoma (RB).
2. Retinoblastoma with at least one eye eligible for conservative management.
3. Patients likely to be compliant with the study requirements and visits, including late follow-up.
4. Patients not previously treated with chemotherapy or radiotherapy for this or any other cancer.
5. Patients with no contraindication to the proposed treatments.
6. Informed consent signed by parents or legal representative.
7. French Social Security System coverage.

Study 1 inclusion criteria:

8.1. Children aged from 6 months to 6 years. 9. Retinoblastoma in at least one eye, deemed manageable with IAC in one side and without IV chemotherapy:

1. Unilateral Retinoblastoma classified as group B, C (if vitreous seeds < 3 mm), D or E with no invasion of the anterior segment, and without massive tumor of more than 2/3 of the eye, eligible for conservative management, or
2. Bilateral Retinoblastoma but with very unbalanced lesions between the two eyes: one eye group D or E without invasion of the anterior segment or massive tumor of more than 2/3 of the eye, eligible for IAC, and the other eye eligible for local treatment only (without IAC).

Study 2 inclusion criteria:

8.2. Retinoblastoma eligible for conservative management although not manageable with IAC:

1. Unilateral Retinoblastoma in children below 6 months of age, classified as Group A, B, C or D, with or without vitreous seeding, compatible with conservative management, or
2. Bilateral Retinoblastoma classified as group A, B, C D, or E without invasion of the anterior segment, and/or massive tumors of more than 2/3 of the eye and eligible for conservative management.

Exclusion Criteria:

Overall study non-inclusion criteria:

1. RB not eligible for conservative management :

   1. Extra-ocular extension of the disease, or
   2. Group E eyes with invasion of the anterior segment, and/or massive tumors of more than 2/3 of the eye.
2. Patient older than 6 years of age.
3. Patients with another associated disease contra indicating systemic chemotherapy.
4. Previously treated retinoblastoma by chemotherapy.
5. Patients already treated for another malignant disease.
6. Patient with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
7. Patients whose parents have not accepted the treatment regimen after explanation of it.
8. Contraindication to study drug mentioned in SmPC (Summary of Products Characteristics) of the study drugs.
9. Inclusion in another experimental anti-cancer drug therapy.

   Study 1 non-inclusion criteria:
10. Any contraindication or concomitant disease that would preclude the Study 1 treatment procedure and could delay treatment.

These patients should be eligible for Study 2.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 225 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2035-01-20 (Estimated); Study Completion 2036-01-20 (Estimated)

PRIMARY OUTCOMES:
Study 1: Rate of eye preservation | 24 months after randomization
  Rate of eye preservation in the 2 treatments' arms
Visual function | when patient is 6 years old and at least 24 months of follow-up after study inclusion
  Percentage of patients with major, mild or no impairment of visual function according to WHO criteria, i.e. normal bilateral visual acuity (≥ 6/10) or mild bilateral visual impairment (3/10 to 5/10) according to tumor location and extension

SECONDARY OUTCOMES:
Ocular toxicity | Up to 24 months after inclusion in the study
  Percentage of patients with at least one grade-3 or -4 toxicity (CTCAE v. 5.0)
Systemic toxicity | Up to 24 months after inclusion in the study
  Rate of specific grade 3-4 toxicity (CTCAE v. 5.0)
Relapse | within 24 months after inclusion
  Percentage of patients with relapse within 24 months after inclusion, broken down into: Local relapse, Extra-ocular relapse
Second malignant tumor | 24 months after study inclusion
  Percentage of patients with second malignant tumor within 24 months after study inclusion
Additional assessment of visual function | In the year patients turn 6 years of age and at least 24 months of treatment
  Additional assessment of visual function at follow-up: Percentage of patients at each of the four levels of visual acuity according to WHO criteria
Retinal assessment | In the year patients turn 6 years of age and at least 24 months of treatment
  Optical Coherence Tomography (OCT) and Optical Coherence Tomography-Angiography (OCT-A) measures on retina
Integration at school | In the year patients turn 6 years of age and at least 24 months of treatment
  Rate of children able to attend the common primary school : without specific help or with the help of a dedicated person and/or with specific features to facilitate reading and writing

CONTACTS AND LOCATIONS:
Overall Officials: Livia LUMBROSO LE ROUIC, MD, Principal Investigator — Institut Curie
Locations (28):
- France (28):
  - La Reunion - Chr Felix Guyon, Saint-Denis, La Réunion
  - Amiens Chu, Amiens
  - Angers Chu, Angers
  - BESANCON CHU Hopital Jean Minjoz, Besançon
  - Bordeaux Chu, Bordeaux
  - BREST CHRU Hopital Morvan, Brest
  - CAEN CHU, Caen
  - CHU ESTAING Centre Régional de Cancérologie et Therapie Cellulaire Pediatrique (CRCTCP), Clermont-Ferrand
  - DIJON CHU Hopital François Mitterand, Dijon
  - Grenoble Chu, Grenoble
  - LILLE Centre Oscar Lambret, Lille
  - Limoges Chu, Limoges
  - LYON Centre Léon Bérard, Lyon
  - Marseille Chu, Marseille
  - MONTPELLIER CHU Hopital Arnaud De Villeneuve, Montpellier
  - NANTES CHU Hopital Mere-Enfant, Nantes
  - NICE CHU Hopital Archet 2, Nice
  - Institut Curie, Paris
  - PARIS Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Poitiers Chu, Poitiers
  - Reims Chu, Reims
  - Rennes Chu, Rennes
  - Rouen Chu, Rouen
  - Saint Etienne Chu, Saint-Etienne
  - Strasbourg Chu, Strasbourg
  - Toulouse Chu, Toulouse
  - TOURS CHU Hopital Clocheville, Tours
  - Nancy Chu, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).